CLINICAL TRIAL: NCT05110404
Title: EFFECT OF HIGH VERSUS LOW-VOLUME HIGH INTENSITY INTERVAL TRAINING ON GLYCEMIC AND LIPIDS CONTROL IN TYPE 2 DIABETES
Brief Title: COMPARISON BETWEEN TWO SUB-TYPES OF HIGH INTENSITY INTERVAL TRAINING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Mohamed Mahmoud Mohamed, physiotherapist holds a master's degree in Physical therapy for Cardiovascular, Respiratory disorders and geriatrics, Faculty of physical therapy, Cairo university., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002900
Record Dates: First submitted 2021-10-21; First posted 2021-11-08 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus
Keywords: DM
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (A): The high-volume HIIT (Active Comparator): Exercise group A (n=30): It will include patients that will perform high-volume high-intensity interval training (HIIT), and will receive medical intervention.
  Interventions: Other: The high-volume HIIT
- Group (B): The low-volume HIIT (Active Comparator): Exercise group B (n=30): will receive medical intervention. that will perform the low-volume high-intensity interval training, and will receive medical intervention.
  Interventions: Other: The low-volume HIIT
- Group C (No Intervention): patients will receive medical intervention only.

INTERVENTIONS:
Other: The high-volume HIIT — patients will undergo a warm up at 65%-70% of HRpeak for 5 minutes, and then they will walk on a treadmill for 4 intervals of 4 min each at an intensity corresponding to 85%-90% of HRpeak with 3 min active recovery interval interval in between at 65%-75% of HRpeak. Finally, a 3-min cool-down period will be permitted. The speed and the inclination of the treadmill will be adjusted between intervals to ensure that all patients are exercising at the desired target heart rate monitored by Pulse Oximeter.
  Arms: Group (A): The high-volume HIIT
Other: The low-volume HIIT — Each session will start with a 5-minute warm up at 65-70% of peak HR. Then they will walk on a treadmill for 4 intervals of 2 min each at an intensity corresponding to 85%-90% of HRpeak with three intervals of active recovery in between for 2 min at 65%-75% of HRpeak. Finally, a 3-min cool-down period will be permitted.
  Arms: Group (B): The low-volume HIIT

SUMMARY:
Recently, HIIT has been recommended by the American diabetes association for type 2 diabetes. The high-volume HIIT has been studied extensively in patients with type 2 diabetes, however, little is known about the effectiveness of low-volume HIIT regarding target glycemic or lipid control in these patients. Therefore, the purpose of this study is to compare between two subtypes of HIIT (i.e. the low-volume HIIT versus the high-volume HIIT) with respect to exercise-induced changes in blood glucose, lipid profile and anthropometry in patients with type 2 diabetes mellitus. Statement of the Problem Is there any difference between the effect of high-volume and the low-volume high intensity interval training on glycemic and lipids control in type 2 diabetes?

Purpose of the study:

To assess the effect of the high-volume versus the low-volume high intensity interval training on glycemic and blood lipids control in type 2 diabetes.

Null Hypothesis:

There will be no difference between the effect of the high-volume versus the low-volume high intensity interval training on glycemic and blood lipids control in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Type II diabetes mellitus diagnosed by a physician as having HbA 1c of > 6.5%.
2. An established diagnosis of T2DM for at least 1year and less than 5 years.
3. Women patients.
4. Age between 35 to 45 years old.
5. Systolic Blood pressure less than or equal 130 mmHg.
6. Obese patients (BMI is between 30 and 39.9 kg/m 2 )
7. Patients with HbA 1c of 7-9%.
8. A self-reported sedentary lifestyle.
9. Patients receiving oral hypoglycemic medications described by the physician
10. Patients with hyperlipidemia.

Exclusion Criteria:

1. Patients with Cardiac diseases.
2. Patients with glaucoma.
3. Patients with diabetic complications (Diabetic foot, retinopathy, nephropathy, and diabetic peripheral neuropathy).
4. Musculoskeletal or neurological limitations to physical exercise.
5. Pregnancy
6. Patients under insulin therapy
7. Patients with poorly controlled DM (HbA1c > 9%)
8. Bronchial asthma and chronic obstructive pulmonary disease.
9. Smokers.
10. Morbidly obese BMI ≥ 40 kg/m 2
11. Males.

11. Systolic Blood pressure more than 130 mmHg. 12. Anemia ( hemoglobin < 12 g/dL) 13. Osteopenia.

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-12-25 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
body mass index | 12 weeks
  change in body mass index
waist circumference | 12 weeks
  change in waist circumference
waist/hip ratio | 12 weeks
  change in waist/hip ratio
Systolic and diastolic blood pressure | 12 weeks
  change in Systolic and diastolic blood pressure
HbA1c | 12 weeks
  change in HbA1c
fasting & 2-h post prandial blood glucose | 12 weeks
  change in fasting & 2-h post prandial blood glucose
fasting lipid profile | 12 weeks
  change in fasting lipid profile

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Ahmad AM, Mahmoud AM, Serry ZH, Mohamed MM, Abd Elghaffar HA. Effects of low-versus high-volume high-intensity interval training on glycemic control and quality of life in obese women with type 2 diabetes. A randomized controlled trial. J Exerc Sci Fit. 2023 Oct;21(4):395-404. doi: 10.1016/j.jesf.2023.08.003. Epub 2023 Aug 30. PMID 37954548